CLINICAL TRIAL: NCT01581411
Title: Phase 1 Trial of Intra-Ophthalmic Artery Thrombolysis for Treating Recent Severe Central Retinal Vein Occlusion
Brief Title: Intra-arterial Thrombolysis for Severe Recent Central Retinal Vein Occlusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRVO-IAT1
Record Dates: First submitted 2012-04-12; First posted 2012-04-20 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Central Retinal Vein Occlusion
Keywords: central retinal vein occlusion; macular edema; vision loss; relative afferent papillary defect
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema; Vision Disorders | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IA t-PA (Experimental): intra-ophthalmic artery injection of tissue plasminogen activator
  Interventions: Drug: Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Tissue Plasminogen Activator — Intra-ophthalmic artery injection of 2 mg t-PA over 10 minutes followed by 10 mg t-PA over 2 hours
  Other Names: intra-arterial thrombolysis

SUMMARY:
Central retinal vein occlusion (CRVO) is a common cause of vision loss, typically affecting individuals during the fifth through seventh decade of life. Eyes with severe CRVO have a poor visual prognosis because current treatments address only secondary complications of CRVO without treating its cause. Intra-ophthalmic artery injection of a small dose of t-PA (clot busting medicine), also called intra-ophthalmic artery thrombolysis, may reopen the central retinal vein-and address the cause of the disease- without exposing the subject to the risks of systemic thrombolysis. Our project aims to evaluate the safety and efficacy of intra-ophthalmic artery thrombolysis in subjects with CRVO.

DETAILED DESCRIPTION:
1. Study hypothesis: Injection of t-PA, a thrombolytic drug (clot busting medicine)into the ophthalmic artery (the blood vessel feeding the eye), in patients with recent severe central retinal vein occlusion, may reopen the central retinal vein and improve retinal blood flow, which may in turn improve visual acuity and prevent the long-term complications of the disease.
2. Experimental intervention: An outpatient procedure during which the ophthalmic artery is selective catheterized (with a small plastic tube called a microcatheter introduced from the artery of the leg) and infused with t-PA during two hours.

ELIGIBILITY:
Inclusion Criteria:

* Severe CRVO diagnosed on

  * presence of relative afferent papillary defect (RAPD)
  * or visual acuity of 20/200 or worse
* Symptom onset within 2 weeks
* Age > 18 years old
* Patient is able and willing to give informed consent

Exclusion Criteria:

* Futile intervention: no light perception, absence of perfusion on fluorescein angiography.
* Contra-indication to thrombolysis: active or recent (1 month) internal bleeding, cerebrovascular accident, major organ surgery, major trauma; intracranial neoplasm or vascular malformation, known bleeding diathesis, severe uncontrolled arterial hypertension, pregnancy (women of childbearing age must have a negative serum pregnancy test), or any other condition which in the opinion of the investigators would preclude the use of thrombolytic agents.
* High-risk catheterization: history of stroke or TIA; carotid bruit or known carotid occlusive disease; any cardiovascular condition that in the opinion of the investigators may increase the risk of catheterization of the ophthalmic artery.
* Ocular criteria: Intraocular neovascularization (secondary to any etiology), vitreous hemorrhage, inflammatory eye disease, any condition that precludes fundus photography or fluorescein angiography.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Improvement of retinal perfusion on the 1-week fluorescein angiogram, with no severe complications. | One week

SECONDARY OUTCOMES:
Number of patients with 3 or more lines of visual acuity improvement during follow up. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Y Pierre Gobin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College/ New York Presbyterian hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No